CLINICAL TRIAL: NCT07064226
Title: Transcultural and Multidimensional Validation of dIgital Rehabilitation Intervention of COgnitive Resources Domain-Oriented - Work Package 4
Brief Title: Validation of a Digital Intervention to Rehabilitate Cognitive Resources
Acronym: MI-RICORDO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Collaborators: Università Carlo Cattaneo , Castellanza (Unknown); ASTIR (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MI-RICORDO; FP-1321 (Other: THCS https://www.thcspartnership.eu/)
Record Dates: First submitted 2025-07-03; First posted 2025-07-14 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Mild Cognitive Impairment (MCI); Subjective Memory Complaint; Dementia Alzheimer Type
Keywords: telerehabilitation; Alzheimer disease; cognitive decline; cognitive rehabilitation; Digital medicine; Dementia; Mild Cognitive Impairment; neuroimaging
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease; Dementia | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Randomized control study with 2 groups: experimental rehabilitation intervention (Ricordo) vs Treatment as usual
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RICORDO (Experimental): Participants will carry out telerehabilitation using a digital platform [http://www.ricordo-dtx.com/], at home, autonomously.
  Interventions: Other: RICORDO
- Treatment as Usual (TAU) (Active Comparator): Participants will follow a traditional paper-and-pencil rehabilitation protocol at home, autonomously.
  Interventions: Other: Treatment as Usual (TAU)

INTERVENTIONS:
Other: RICORDO — During the RICORDO intervention, participants will engage in a multidomain cognitive telerehabilitation program using a digital platform ([http://www.ricordo-dtx.com/]), which allows for personalized interventions through an adaptive algorithm allowing an increment in task difficulties according to patients' needs. The treatment can be self-administered by the patient at home. The program lasts five weeks, with three treatment sessions per week, each lasting approximately 45 minutes.
  The active control group (TAU) will undergo the same type of treatment with the following differences: the digital platform will not be used, as the treatment will consist solely of paper-and-pencil exercises; and there will be no personalization of the exercises, since automatic adaptation is not possible.
  Arms: RICORDO
Other: Treatment as Usual (TAU) — As described above, this type of intervention will consist in a multidomain cognitive rehabilitation treatment to be self administered by the participants at home with pencil paper excercises. Treatment will last 5 weeks, 3 sessions per week, each lasting approximately 45 minutes. The treatment will follow a predefined incremental difficulty structure since no personalization is available.
  Arms: Treatment as Usual (TAU)

SUMMARY:
The goal of this clinical trial is to learn if the use of a digital cognitive rehabilitation system named RICORDO, that is flexible and capable of adapting the rehabilitation pathway according to the needs and capacity of the patients will prove effective for subjects with Subjective Memory Complaint or with Mild Cognitive Impairment or with Mild Dementia.

The main questions it aims to answer are:

Will the RICORDO rehabilitation treatment, lead to an improvement in the global cognitive level? Will the RICORDO rehabilitation treatment lead to improved activation of participants in managing their own health and healthcare? Researchers will compare the multidomain cognitive rehabilitation strategy of RICORDO digital solution, with a standard paper pencil rehabilitation care (usual care).

Participants will undergo a comprehensive neuropsychological evaluation immediately before, immediately after and six months after the completion of the rehabilitation program.

Both interventions, the experimental and the usual care, will last 5 weeks, with 3 weekly sessions of 45 minutes each and can be done autonomously by the patient at home.

ELIGIBILITY:
Inclusion Criteria:

1. Montreal Cognitive Assessment (MoCA) score > 17.79;
2. Clinical Dementia Rating (CDR) Scale score ≤ 1;
3. Education level > 3 years;
4. Age ≥ 65 years;
5. Informed consent to participate, confirmed by signing the consent form;
6. Availability of a caregiver/study partner able to support the participant;
7. Stable pharmacological treatment (past 3 months) with acetylcholinesterase inhibitors, if applicable.

Exclusion criteria:

1. Presence of dysmetria or marked auditory/visual or communication disorders preventing the participation to the trial;
2. Presence of ongoing rehabilitation program at the time of enrollment or in the 3 months prior to enrollment;

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2025-09-10 (Estimated); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in global cognitive functioning and subdomains measured by Montreal Cognitive Assessment MoCA | Baseline, after 5 weeks (End of treatment), 6 months after baseline (Follow-up)
  MoCA is a screening test for cognitive deficits. It measures the global cognitive functioning and includes several tasks involving different domains: visuospatial/executive function, language, selective and sustained attention, abstraction, memory and orientation. Score ranges from 0 to 30 with higher scores indicating better general cognitive performance.
Change in Activation level of Patients measured by Patient Activation Measure 13 (PAM13) | Baseline, after 5 weeks (End of treatment), 6 months after baseline (Follow-up)
  The Patient Activation Measure (PAM-13) is a 13-item instrument designed to evaluate an individual's knowledge, skills, and confidence in effectively managing their health and healthcare. The total PAM-13 score ranges from 0 to 100, with higher scores indicating greater levels of activation and more favorable outcomes. Individuals classified in the lowest activation level typically lack awareness of their role in managing their health, demonstrate limited health-related knowledge, and possess underdeveloped self-management abilities. In contrast, those in the highest activation level exhibit proactive health behaviors, possess well-established self-management competencies, and demonstrate resilience in response to stress or health-related changes.

SECONDARY OUTCOMES:
Change in memory in everyday situations measured by Everyday Memory Questionnaire Revised | Baseline, after 5 weeks (End of treatment), 6 months after baseline (Follow-up)
  The Everyday Memory Questionnaire (EMQ) is a self-report instrument designed to assess subjective experiences of memory failure in daily life. The revised version comprises 13 items, each describing a specific memory-related situation. Respondents rate the frequency with which they experience each situation using a 5-point Likert scale. The total score is calculated as the sum of all item responses and ranges from 0 to 52, with higher scores indicating a greater frequency of everyday memory lapses.
Change in depressive symptoms measured by Beck Depression Inventory II | Baseline, after 5 weeks (End of treatment), 6 months after baseline (Follow-up)
  The Beck Depression Inventory II is a self report questionnaire to evaluate the depression level. It consists of 21 questions, each scored on a 4-point scale, with a total score ranging from 0 to 63. The total score is calculated by summing the responses to all 21 questions. HIgher scores indicate more severe deflection of mood tone. The BDI-II can be used to assess the effectiveness of treatment interventions.
Change in mood measured by Positive and Negative Affect Scale (PANAS) | Baseline, after 5 weeks (End of treatment), 6 months after baseline (Follow-up)
  The Positive and Negative Affect Schedule (PANAS) is a self-administered questionnaire designed to assess affective states. It consists of two distinct subscales that measure positive affect (PA) and negative affect (NA), respectively. Each subscale comprises ten descriptive adjectives, with participants rating the extent to which they have experienced each emotion on a 5-point Likert scale, ranging from 1 (very slightly or not at all) to 5 (extremely). The overall PANAS score is calculated by summing the ratings for the items within each subscale, yielding separate PA and NA scores. Score ranges from 10 to 50. Higher scores on each subscale reflect greater intensity of the corresponding affect. In scoring, values from the positive affect items contribute to the PA score, while values from the negative affect items contribute to the NA score.
Change in anxiety level measured by State-Trait Anxiety Inventory (STAI- Y state) | Baseline, after 5 weeks (End of treatment), 6 months after baseline (Follow-up)
  The STAI-Y is a frequeltly used self-reported questionnaire to measure state anxiety (20 items). Each item is rated on a 4-point scale (from "Almost Never" to "Almost Always"). STAI is scored by summing ratings for each item (range 0-80). Higher scores indicate greater anxiety.
Change in Language and Executive Functions evaluated by Phonemic/Semantic alternate fluency test | Baseline, after 5 weeks (End of treatment), 6 months after baseline (Follow-up)
  The Phonemic/Semantic Alternate Fluency Test (Costa et al., 2014) is a verbal fluency task designed to assess executive functioning, particularly cognitive flexibility and lexical access. Participants are required to alternately generate words beginning with a specific letter (phonemic fluency) and belonging to a specific semantic category (semantic fluency) within a limited time frame. This alternating condition increases task complexity and places greater demands on mental set shifting compared to traditional fluency tasks.
Change in visuospatial abilities evaluated by Benson Figure Copy and recall | Baseline, after 5 weeks (End of treatment), 6 months after baseline (Follow-up)
  The Benson Figure Test is a neuropsychological assessment used to evaluate visuospatial abilities, visual memory, and constructional skills. Patients are asked to copy a complex figure and to recall it after 10 minutes.
Change in visuoperceptual and attentional abilities measured by Trail Making Test (TMT parts A and B) | Baseline, after 5 weeks (End of treatment), 6 months after baseline (Follow-up)
  The Trail Making Test (TMT) is a neuropsychological test used to assess attention, mental flexibility, and motor coordination. It involves connecting a sequence of targets (numbers or alternating numbers and letters) as quickly as possible, while maintaining accuracy. The test has two parts, A and B, with Part B requiring a switch in task requirements. The scoring of TMT consists in the time used to complete each part of the test. Higher execution times indicate poorer performance.
Change in patient's self-rated health measured by EuroQol five dimensions (5D) and five levels (5L) | Baseline, after 5 weeks (End of treatment), 6 months after baseline (Follow-up)
  The EQ-5D-5L is a standardized measure of health status, consisting of two parts: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The descriptive system evaluates five dimensions of health: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has five response levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. The EQ VAS captures the patient's self-rated health on a vertical visual analogue scale, with endpoints labeled 'The best health you can imagine' (scored as 100) and 'The worst health you can imagine' (scored as 0).
Change in immediate recall memory measured by the Free and Cued Selective Reminding Test (FCSRT) | Baseline, after 5 weeks (End of treatment), 6 months after baseline (Follow-up)
  The patient is instructed to freely and cuedly recall as many items as possible. The score corresponds to the total number of recalled items across the three immediate trials (range: 0-36). Higher scores indicate greater memory performance.
Change in delayed recall memory measured by the Free and Cued Selective Reminding Test (FCSRT) | Baseline, after 5 weeks (End of treatment), 6 months after baseline (Follow-up)
  The patient is asked to recall as many items as possibile after 30 min from learning phase. The score corresponds to the number of recalled items across the three trials (range: 0-12).
Change in Theory of Mind ability evaluated by Yoni-48 task | Baseline, after 5 weeks (End of treatment), 6 months after baseline (Follow-up)
  The Yoni-48 task is a computerized measure of Theory of Mind (ToM), specifically designed to assess first- and second-order affective and cognitive mentalizing. It consists of 48 visual stimuli presented on a computer screen, where a cartoon character named "Yoni" is shown with four surrounding elements. The mentalizing stimuli comprise 21 affective and 21 cognitive ToM items and are divided into 16 first-order (8 affective, 8 cognitive) and 26 second-order (13 affective and 13 cognitive) ToM stimuli. the remaining 6 are non mentalizing - control items. The scores are summed and adjusted for demographics to compute an accuracy index ranging from 0 (poorer performance) to 1 (better performance).

OTHER OUTCOMES:
Changes in Fractional Anisotropy (FA) and Mean Diffusivity (MD) as detected by Diffusion Weighted Magnetic Resonance Imaging (DWI). | Baseline, after 5 weeks (End of treatment), 6 months after baseline (Follow-up)
  DWI sequences will be collected to detect changes in FA and MD (these indices are complementary and need to be considered together to be interpreted) to evaluate structural connectivity.
Changes in Functional Connectivity (FC) as detected by resting state functional Magnetic Resonance Imaging (rs-fMRI) | Baseline, after 5 weeks (End of treatment), 6 months after baseline (Follow-up)
  Resting-State fMRI (Multi echo - Multi-Band) images will be collected for the assessment of the FC before and after intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Valeria Blasi, Medical Doctor, Principal Investigator — IRCCS Fondazione Don Carlo Gnocchi ONLUS
Locations (1):
- IRCCS Fondazione Don Carlo Gnocchi ONLUS; Center of Advance Diagnostic and Therapy ( CADiTeR), Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Spielberger CD, Gorsuch RL, Lushene RE, et al. State-Trait Anxiety Inventory for adults: manual, instrument and scoring guide. Palo Alto: Mind Garden; 1983
- [Background] BECK AT, WARD CH, MENDELSON M, MOCK J, ERBAUGH J. An inventory for measuring depression. Arch Gen Psychiatry. 1961 Jun;4:561-71. doi: 10.1001/archpsyc.1961.01710120031004. No abstract available. PMID 13688369
- [Background] Morris JC. The Clinical Dementia Rating (CDR): current version and scoring rules. Neurology. 1993 Nov;43(11):2412-4. doi: 10.1212/wnl.43.11.2412-a. No abstract available. PMID 8232972
- [Background] Balestroni G, Bertolotti G. [EuroQol-5D (EQ-5D): an instrument for measuring quality of life]. Monaldi Arch Chest Dis. 2012 Sep;78(3):155-9. doi: 10.4081/monaldi.2012.121. Italian. PMID 23614330
- [Background] Isernia S, Rossetto F, Shamay-Tsoory S, Marchetti A, Baglio F. Standardization and normative data of the 48-item Yoni short version for the assessment of theory of mind in typical and atypical conditions. Front Aging Neurosci. 2023 Jan 12;14:1048599. doi: 10.3389/fnagi.2022.1048599. eCollection 2022. PMID 36711213
- [Background] Possin KL, Laluz VR, Alcantar OZ, Miller BL, Kramer JH. Distinct neuroanatomical substrates and cognitive mechanisms of figure copy performance in Alzheimer's disease and behavioral variant frontotemporal dementia. Neuropsychologia. 2011 Jan;49(1):43-8. doi: 10.1016/j.neuropsychologia.2010.10.026. Epub 2010 Oct 26. PMID 21029744
- [Background] Costa A, Bagoj E, Monaco M, Zabberoni S, De Rosa S, Papantonio AM, Mundi C, Caltagirone C, Carlesimo GA. Standardization and normative data obtained in the Italian population for a new verbal fluency instrument, the phonemic/semantic alternate fluency test. Neurol Sci. 2014 Mar;35(3):365-72. doi: 10.1007/s10072-013-1520-8. Epub 2013 Aug 21. PMID 23963806
- [Background] Giovagnoli AR, Del Pesce M, Mascheroni S, Simoncelli M, Laiacona M, Capitani E. Trail making test: normative values from 287 normal adult controls. Ital J Neurol Sci. 1996 Aug;17(4):305-9. doi: 10.1007/BF01997792. PMID 8915764
- [Background] Frasson P, Ghiretti R, Catricala E, Pomati S, Marcone A, Parisi L, Rossini PM, Cappa SF, Mariani C, Vanacore N, Clerici F. Free and Cued Selective Reminding Test: an Italian normative study. Neurol Sci. 2011 Dec;32(6):1057-62. doi: 10.1007/s10072-011-0607-3. Epub 2011 May 19. PMID 21594655
- [Background] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- [Background] Royle J, Lincoln NB. The Everyday Memory Questionnaire-revised: development of a 13-item scale. Disabil Rehabil. 2008;30(2):114-21. doi: 10.1080/09638280701223876. PMID 17852284
- [Background] Hibbard JH, Stockard J, Mahoney ER, Tusler M. Development of the Patient Activation Measure (PAM): conceptualizing and measuring activation in patients and consumers. Health Serv Res. 2004 Aug;39(4 Pt 1):1005-26. doi: 10.1111/j.1475-6773.2004.00269.x. PMID 15230939
- [Background] Dapor C, Devita M, Iannizzi P, Arbia E, Bruzzano A, Dessi M, Lupi D, Rolandino GM, Rossi M, Saccomano A, Siccardi E, Simonetto A, Vuerich G, Zuliani S, Priftis K. The Montreal cognitive assessment (MoCA) 8.1 version, including the memory index score (MoCA-MIS): Italian norms. Neurol Sci. 2025 Jun;46(6):2581-2589. doi: 10.1007/s10072-025-08066-1. Epub 2025 Mar 17. PMID 40095163
- [Derived] Blasi V, Isernia S, Rossetto F, Pagliari C, Borgnis F, Pirastru A, Marzulli M, Foglia E, Garagiola E, Baglio F. Study protocol for a randomized controlled trial assessing clinical efficacy of digital cognitive rehabilitation for preclinical and mild clinical stages of alzheimer's disease continuum: the MI-RICORDO project. BMC Psychiatry. 2025 Nov 11;25(1):1075. doi: 10.1186/s12888-025-07531-7. PMID 41219714